CLINICAL TRIAL: NCT02538471
Title: LY2157299 Monohydrate (LY2157299) and Radiotherapy in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of patient accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1505016222
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Radiation; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 - Study Drug & Radiation therapy (Experimental): Study Drug: Enrolled patients will receive 300 mg/day of LY2157299. LY2157299 will be administered as an oral drug tablet.
  The study drug will be administered orally on a 28-day cycle (1 cycle=28 days), every 2 weeks, or 14 days on / 14 days off. Blood samples will be obtained at baseline, and weeks 2, 6 and 15 for immune monitoring.
  Radiation therapy : Patients will receive Radiation therapy to a metastatic site at a dose of 7.5 Gy, given consecutively on days 1, 3 and 5, during Week 1 of their treatment.
  Interventions: Radiation: Radiation therapy; Drug: Study Drug

INTERVENTIONS:
Radiation: Radiation therapy — Imaging by PET/CT will be performed at baseline, 5 weeks and 15 weeks. The chosen metastatic sites will receive conformal external beam radiation 7.5 Gy/fraction x 3, to a total of 22.5 Gy over the course of one week.
  Other Names: Radiation
Drug: Study Drug — Patients will receive 300 mg/day of study drug administered via oral drug tablet every day for 14 days on and 14 days off (=28 day cycle) .
  Other Names: Study Drug - oral

SUMMARY:
Patients with metastatic breast cancer receiving at least one single agent chemotherapy and demonstrating stable disease or disease progression at two consecutive clinical/radiological assessments (at an interval of at least 2 weeks).

Transforming growth factor-beta (TGFΒ) blockade will enhance response of irradiated tumors and improve the function of Dendritic and T cells. Patients will receive 300 mg/day of study drug administered via oral drug tablet every day for 14 days on and 14 days off (=28 day cycle). Radiation to a metastatic site will be delivered at a dose of 7.5 Gy, given consecutively on days 1-3-5.

DETAILED DESCRIPTION:
Transforming growth factor-beta (TGFβ) is a pleiotropic cytokine which belongs to a superfamily of ligands, including bone morphogenetic proteins and activins [1-5]. Under normal conditions, members of the TGFβ family maintain homeostasis in many organ systems. In normal and non-cancerous cells, TGFβ limits the growth of epithelial, endothelial, neuronal, and hematopoietic cell lineages through anti-proliferative and apoptotic responses. In addition, TGFβ exerts potent effects that influence immune function, cell proliferation/ functional differentiation, cell adhesion, extracellular matrix production, cell motility, angiogenesis, and cytokine production. TGFβ has been implicated as an important factor in the growth, progression, and metastatic potential of advanced cancers. Although TGFβ has been shown to suppress the growth of epithelial cells in the early stages of tumor development (premalignant conditions), the effect on advanced cancers is more complex [1, 5-6]. Increased production of TGFβ has been found in many neoplasms such as breast, prostate, gastric, renal, and epidermal carcinomas, and elevated plasma TGFβ levels in patients have been correlated with advanced disease, metastases, and lower survival rates [7-13]. In these later stage cancers, TGFβ induced growth suppression is lost, and instead, TGFβ promotes tumor growth and metastasis.

Eli Lilly has developed and produced a Transforming Growth Factor-beta (TGF-β) receptor type-1 kinase inhibitor. LY2157299 monohydrate (LY2157299) is a small molecule that inhibits the TGF-β receptor type 1 kinase activity. LY2157299 was developed to investigate its activity in patients with glioblastoma where TGF-β has been demonstrated to play a specific role in tumor progression. In addition, LY2157299 was investigated in other patient populations, either as a stand-alone therapy or in combination with standard anti-tumor treatment regimens for indications including hepatocellular carcinoma and pancreatic cancer. Future investigations include indications with likely TGF-β associated pathway activation, such as melanoma, breast and prostate cancer as well as hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria :

1. Biopsy proven breast carcinoma which is persistent and metastatic or recurrent and metastatic.
2. Patients must have failed at least one line of chemotherapy for metastatic disease.
3. Patients who are Human epidermal growth factor 2 +(HER2+) as defined by American Society of Clinical Oncology and College of American Pathologists (ASCO CAP) guidelines must have failed all prior therapy known to confer clinical benefit
4. Patients must have at least 3 distinct metastatic sites with at least one measurable lesion which is at least 1 cm or larger in largest diameter
5. At the time of enrollment, patients must be ≥ 4 weeks since all of the following treatments (and recovered from the toxicity of prior treatment to <= Grade 1, exclusive of alopecia):

   major surgery; radiotherapy; chemotherapy (note: must be ≥ 6 weeks since therapy if treated with a nitrosourea, mitomycin, or monoclonal antibodies such as bevacizumab); immunotherapy; Biotherapy/targeted therapies.
6. Patient ≥ 18 years of age. Patient life expectancy > 6 months. Eastern cooperative group (ECOG) of 0 or 1
7. Adequate organ function including:

   1. Marrow: Hemoglobin >= 10.0 g/dL, absolute neutrophil count (ANC) >=1,500/mm3, and platelets >=100,000/mm3.
   2. Hepatic: Serum total bilirubin <=1.5 x upper limit of normal (ULN) (Patients with Gilbert's Disease may be included if their total bilirubin is <= 3.0 mg/dL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 2.5 x ULN. If the patient has known liver metastases, an ALT and/or AST <= 5 x ULN are allowed.
   3. Renal: Estimated or measured creatinine clearance >= 60 mL/min.
   4. Other: Prothrombin time (PT) and partial thromboplastin time (PTT) < ULN.
8. Patients must have negative tests (antibody and/or antigen) for hepatitis viruses B and C unless the result is consistent with prior vaccination or prior infection with full recovery.
9. Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment.

Exclusion Criteria :

1. Patients diagnosed with another malignancy - unless following curative intent therapy, the patient has been disease free for at least 2 years and the probability of recurrence of the prior malignancy is < 5%. Patients with curatively treated early-stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study.
2. Concurrent cancer therapy is not permitted.
3. Uncontrolled central nervous system (CNS) metastases, meningeal carcinomatosis, malignant seizures, or a disease that either causes or threatens neurologic compromise (e.g., unstable vertebral metastases).
4. History of ascites or pleural effusions, unless successfully treated.
5. Patients with an organ transplant, including those that have received an allogeneic bone marrow transplant.
6. Patients on immunosuppressive therapy including:

   1. Systemic corticosteroid therapy for any reason, including replacement therapy for hypoadrenalism. Patients receiving inhaled or topical corticosteroids may participate (if therapy is < 5 days and is limited to systemic steroids as antiemetics).
   2. Patients receiving cyclosporine A, tacrolimus, or sirolimus are not eligible for this study.
7. Use of investigational agents within 4 weeks prior to study enrollment (within 6 weeks if the treatment was with a long-acting agent such as a monoclonal antibody).
8. Patients with moderate or severe cardiac disease:

   1. have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension.
   2. have documented major electrocardiogram (ECG) abnormalities (not responding to medical treatments) at the investigator's discretion (for example, symptomatic or sustained atrial or ventricular arrhythmias, second- or third-degree atrio ventricular block, complete bundle branch block, ventricular hypertrophy, or recent myocardial infarction).
   3. have major abnormalities documented by echocardiography (ECHO) with Doppler (for example, moderate or severe heart valve function defect and/or left ventricular ejection fraction <50%, evaluation based on the institutional lower limit of normal). For additional details, refer to ECHO protocol.
   4. have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan-Syndrome, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by computed tomography (CT) scan with contrast).
9. B-type Natriuretic Peptide (BNP) above 3 times the baseline value and above the ULN that is sustained consecutive, scheduled blood draws. Troponin I above ULN, high sensitive C-reactive protein (hsCRP) above ULN or Cystatin above ULN.
10. Patients with a remote history of asthma or active mild asthma may participate.
11. Active infection, including unexplained fever (temperature > 38.5 deg.C).
12. Systemic autoimmune disease (e.g., systemic lupus erythematosus, active rheumatoid arthritis, Marfan Syndrome, etc.).
13. A known allergy to any component of LY2157299.
14. Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems include, but are not limited to:

    1. Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy or significantly increase the risk of Serious Adverse Events (SAEs).
    2. Any condition, psychiatric, substance abuse, or otherwise, that, in the opinion of the Investigator, would preclude informed consent, consistent follow-up, or compliance with any aspect of the study
15. Pregnant or nursing women, due to the unknown effects ofLY2157299 on the developing fetus or newborn infant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Study Drug & Radiation Therapy: Study Drug: Enrolled patients will receive 300 mg/day of LY2157299. LY2157299 will be administered as an oral drug tablet.
  The study drug will be administered orally on a 28-day cycle (1 cycle=28 days), every 2 weeks, or 14 days on / 14 days off. Blood samples will be obtained at baseline, and weeks 2, 6 and 15 for immune monitoring.
  Radiation therapy : Patients will receive Radiation therapy to a metastatic site at a dose of 7.5 Gy, given consecutively on days 1, 3 and 5, during Week 1 of their treatment.
  Radiation therapy: Imaging by PET/CT will be performed at baseline, 5 weeks and 15 weeks. The chosen metastatic sites will receive conformal external beam radiation 7.5 Gy/fraction x 3, to a total of 22.5 Gy over the course of one week.
  Study Drug: Patients will receive 300 mg/day of study drug administered via oral drug tablet every day for 14 days on and 14 days off (=28 day cycle) .
Period: Overall Study
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Started | 3
Completed | 1
Not Completed | 2
Not completed — Progression of disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 61 [60 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Patients who have received at least one 14 days cycle of the study drug will be followed for toxicity (lack of grade 4 toxicity- primary safety end point). Physical exam (including labs) will be performed every 2 weeks while on the study. Patients will be followed with follow-up visits monthly for the first three months after completing therapy then annually for 5 years. Adverse Events will be monitored throughout the course of the study using the NCI CTCAE vers. 4.0.
Time Frame: until end of study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Number of Participants Non-irradiated Tumor Lesions That Had a Response.
Description: To determine if treatment with TGFΒ receptor I kinase inhibitor LY2157299 and localized RT achieves an abscopal tumor regression
Time Frame: Until next progression up to 3 years
Population: Only 1 patient completed protocol therapy. 2 patients were removed from the study for disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Number of Participants Who Received Radiation to the Tumor Who Had a Response.
Description: to estimate the local response rate of combining TGFΒ receptor I kinase inhibitor LY2157299 and local radiotherapy
Time Frame: 25 weeks
Population: Only one patient continued past 25 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Number of Participants Who Had a Change in Their T Regulatory Cell Numbers and Function Over the Course of the Study.
Description: To determine if treatment with TGFβ receptor I kinase inhibitor LY2157299 and localized RT alters the numbers and function of T-reg cells in patients with metastatic breast cancer
Time Frame: 2 years
Population: Due to early termination of the study, blood samples at all time points could not be collected. So this outcome measure couldn't be analyzed.
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Enhanced Tumor Specific Immunity.
Time Frame: 2 years
Population: as for outcome 4
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be collected throughout the course of the study up to 3 years.
Description: Adverse events are collected at every study visit.
Arm/Group | Arm 1 - Study Drug & Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Study Drug & Radiation Therapy (N=3)
Intertrochanteric Fracture and Parietal mass and edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia - Grade 3 (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Study Drug & Radiation Therapy (N=3)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Bloating - Grade 1 (Gastrointestinal disorders) | 1 (1)
Musculoskeletal Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of breath - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Hip Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02538471/Prot_SAP_000.pdf